CLINICAL TRIAL: NCT02071355
Title: Phase I, Open Label Study to Examine the Pharmacokinetics, Safety and Tolerability of TMC435 Following Multiple Oral Doses of 100 and 150 mg q.d. in Healthy Chinese Subjects
Brief Title: A Study to Examine the Pharmacokinetics, Safety and Tolerability of Multiple Oral Doses of TMC435 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018526; TMC435HPC1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-02-24; First posted 2014-02-25 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy; Chinese participants; TMC435; Multiple oral doses; Pharmacokinetics; Safety; Tolerability
MeSH Terms: interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Participants will receive 100 mg TMC435 once daily for 7 days.
  Interventions: Drug: TMC435 100 mg
- Group 2 (Experimental): Participants will receive 150 mg TMC435 once daily for 7 days.
  Interventions: Drug: TMC435 150 mg

INTERVENTIONS:
Drug: TMC435 100 mg — Participants will receive TMC435 100 mg capsule once daily from Day 1 to Day 7 after food.
  Arms: Group 1
Drug: TMC435 150 mg — Participants will receive TMC435 150 mg capsule once daily from Day 1 to Day 7 after food.
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine the pharmacokinetics (what the body does to a medication) of TMC435 after multiple oral doses of 100 and 150 mg TMC435 once daily for 7 days in healthy Chinese participants.

DETAILED DESCRIPTION:
This is an open-label (both [participants and investigator] know what treatment participants will receive) and randomized (study medication is assigned by chance) study. The study consists of 3 phases: a screening phase (within 21 days prior to administration of study medication), a treatment phase (from day -1 [1 days before the administration of study medication] to Day 10 including pharmacokinetics sample collection), and follow-up phase (up to 16 days after the last dose of study medication or after dropout [other than withdrawal of consent]). Approximately 32 healthy participants will be equally divided into 2 groups (Group 1 and Group 2) to receive TMC435 for 7 days. Safety will be evaluated by the assessment of adverse events, clinical laboratory tests, vital signs, and physical examination which will be monitored at various timepoints throughout the study. The total duration of study participation for each participant will be approximately 47 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese participants on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram, and clinical laboratory tests performed at screening
* Must be non-smoking for at least 3 months prior to screening as confirmed by a urine cotinine test
* A Body Mass Index (BMI) of 18.0 to 30.0 kg/square meter, extremes included (BMI is calculated as BMI = body weight in kg divided by the square of height in meters)
* Participants must agree to use one of the contraception methods defined in the protocol

Exclusion Criteria:

* Positive human immunodeficiency virus - type 1 and 2; syphilis; hepatitis A, B or C infection at screening
* History or presence of liver or renal clearance insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* History or evidence of current use of alcohol, barbiturate, amphetamine, recreational or narcotic medicines use
* Any history of significant skin disease such as but not limited to, rash or eruptions, allergies, dermatitis, eczema (inflammation of the skin), psoriasis (an inflammatory skin disease), or urticarial (a raised and itchy rash that appears on the skin)
* Female participants who are breastfeeding at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Predose plasma concentration of TMC435 | Predose on Days 1, 5, 6, and 7
Minimum plasma concentration of TMC435 | Postdose on Day 7 (1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours)
Maximum plasma concentration of TMC435 | Postdose on Day 7 (1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours)
Time to reach the maximum plasma concentration of TMC435 | Postdose on Day 7 (1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours)
Area under the plasma concentration-time curve of TMC435 from time of administration up to 24 hours after dosing | Postdose on Day 7 (1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours)
Area under the plasma concentration-time curve of TMC435 from time of administration up to the last time point with a measurable concentration after dosing | Postdose on Day 7 (1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours)
Average steady-state plasma concentration of TMC435 | Postdose on Day 7 (1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours)
Fluctuation index of TMC435 | Postdose on Day 7 (1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours)
  Fluctuation index, ie, percentage fluctuation: variation between maximum (Cmax) and minimum (Cmin) plasma concentration at steady-state, calculated as: 100 x ([Cmax-Cmin]/Css,av). Css,av is an average steady-state plasma concentration.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 47 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Beijing, China